CLINICAL TRIAL: NCT00292084
Title: A Phase II, Multi-Center, Extension Study to Evaluate the Safety and Efficacy of Celgosivir in Combination With Peginterferon Alfa-2b, With or Without Ribavirin, for an Additional 36 Weeks
Brief Title: An Extension Study to Evaluate the Safety and Efficacy of Celgosivir and Peginterferon Alfa-2b, With or Without Ribavirin, in Patients With Chronic Hepatitis C Genotype 1 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioWest Therapeutics Inc (Industry)
Responsible Party: Jim Pankovich, MIGENIX Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV-05-004
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2008-01-21 (Estimated); Status verified 2008-01

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; Celgosivir; HCV; Genotype 1; Non-responders; End of Treatment Response; Sustained Viral Response
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — celgosivir

INTERVENTIONS:
Drug: Celgosivir

SUMMARY:
This is an extension study of HCV-05-002. The objective of this study is to evaluate the safety and efficacy of celgosivir plus peginterferon alfa-2b, with or without ribavirin, for an additional 36 weeks in patients with chronic hepatitis C genotype 1 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed HCV-05-002 only
* 18-65 years of age, inclusive
* Primary diagnosis of chronic HCV infection
* Non-responders to previous pegylated interferon-based therapy

Exclusion Criteria:

* Patients naive to interferon-based therapy for chronic HCV infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-02; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Safety analysis
HCV viral load reduction from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jim Pankovich, Study Director — BioWest Therapeutics Inc
Locations (1):
- Halifax, Nova Scotia, Canada